CLINICAL TRIAL: NCT07113080
Title: The Effect of Lemongrass and Lavender Aromatherapy on Dental Anxiety and Pain Perception in Children Undergoing Local Anesthetic Administration: A Randomized Clinical Trial
Brief Title: Assessing the Efficacy of Lemongrass and Lavender Aromatherapy in Reducing Dental Anxiety and Pain Associated With Local Anesthetic Injections in Pediatric Dental Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hiba Ahmed Eltayeb (Other)
Responsible Party: Sponsor-Investigator, Hiba Ahmed Eltayeb, master degree candidate, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PED-24-13M
Record Dates: First submitted 2025-05-05; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-05

CONDITIONS: Dental Fear and Anxiety
Keywords: aromatherapy; cortisol; dental anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: participants will be randomly assigned into lavender, lemongrass or the control group in which they will be receiving lavender aromatherapy, lemongrass aromatherapy or no intervention respectively
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lavender aromatherapy (Active Comparator): participants in this arm will receive lavender aromatherapy before local anesthesia administration
  Interventions: Drug: lavender essential oil inhaled using face mask
- lemongrass aromatherapy (Active Comparator): participants in this arm will receive lemongrass aromatherapy before the local anesthesia administration
  Interventions: Drug: lemongrass essential oil inhaled using face mask
- control (No Intervention): participants in this arm will not receive any aromatherapy before the local anesthesia administration

INTERVENTIONS:
Drug: lavender essential oil inhaled using face mask — participants will inhale lavender essential oil via nebulizer before local anesthesia administration
  Arms: lavender aromatherapy
Drug: lemongrass essential oil inhaled using face mask — participants will inhale lemongrass essential oil via nebulizer before the local anesthesia administration
  Arms: lemongrass aromatherapy

SUMMARY:
The goal of this clinical trial is to evaluate whether aromatherapy using lemongrass or lavender essential oils can reduce dental anxiety and pain perception in children aged 7-11 years undergoing local anesthetic administration in a pediatric dental setting.

The main questions it aims to answer are:

Does lemongrass or lavender aromatherapy reduce anxiety levels, as measured by salivary cortisol, in children receiving local anesthesia?

Does aromatherapy influence pain perception and physiological stress (heart rate) during the procedure?

Researchers will compare a lavender aromatherapy group, a lemongrass aromatherapy group, and a control group without aromatherapy to see if the essential oils have a calming effect that reduces anxiety and pain compared to no intervention.

Participants will:

Inhale either lavender, lemongrass, or no essential oil (control) for two minutes via nebulizer.

Undergo local anesthesia administration for a dental procedure.

Provide unstimulated and stimulated saliva samples before and after the procedure for cortisol analysis.

Report their pain level using the Wong-Baker Faces Pain Rating Scale.

Have their heart rate measured before and after the procedure using a finger-type pulse oximeter.

DETAILED DESCRIPTION:
Dental anxiety is a common behavioral challenge in pediatric dentistry and can significantly influence the quality of dental care, potentially leading to avoidance of necessary treatments. One of the most anxiety-inducing procedures is the administration of local anesthesia. Excessive fear and pain perception can negatively impact the child's dental experience and long-term oral health behavior.

Aromatherapy, a non-pharmacological method utilizing essential oils from plants, has shown potential in reducing anxiety and promoting relaxation. Lavender essential oil (Lavandula angustifolia) has been extensively studied for its calming and anxiolytic properties in children and adults. Lemongrass (Cymbopogon citratus) also contains bioactive compounds believed to have similar relaxing effects, though its use in pediatric dental settings has not been adequately evaluated.

This randomized clinical trial aims to investigate the effects of lavender and lemongrass aromatherapy on anxiety levels and pain perception in children aged 7-11 years undergoing local anesthetic administration at the pediatric dentistry department, Faculty of Dentistry, Ain Shams University.

Forty-eight medically free children, with no prior dental visits and who fall within Frankl behavioral rating scale levels 3 or 4, will be randomly assigned to one of three groups:

Lavender aromatherapy group

Lemongrass aromatherapy group

Control group (no aromatherapy)

Children in the intervention groups will inhale either lavender or lemongrass essential oil via a nebulizer for 2 minutes prior to receiving local anesthesia. The control group will receive standard care with no aromatherapy. All local anesthetic injections will be performed using 4% articaine with 1:100,000 epinephrine after applying topical anesthesia to dry mucosa.

To objectively assess anxiety levels, salivary cortisol will be collected before and after the procedure using an unstimulated/stimulated saliva method. Cortisol concentrations will be analyzed using a commercial ELISA kit. Pain perception will be evaluated immediately after the procedure using the Wong-Baker Faces Pain Rating Scale - a validated self-reported tool for children. Heart rate will also be recorded before and after treatment using a finger-type pulse oximeter as a physiological stress marker.

The primary objective is to determine whether either essential oil significantly reduces anxiety levels, as evidenced by changes in salivary cortisol. Secondary outcomes include differences in reported pain and heart rate between groups. The study uses simple randomization with opaque envelope allocation concealment and blinding of outcome assessors (statistician and lab technician). Due to the nature of the intervention, operator and participant blinding is not possible.

This study may offer a practical, non-invasive adjunctive method to manage dental anxiety and pain in children, improving patient cooperation and long-term dental health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* children aged 7-11 years
* medically free
* children category 3 or 4 according to Frankle behavior rating scale
* patients who approve of signing informed consent and give child assent
* children with at least one vital primary molar with deep carious lesion

Exclusion Criteria:

* children with a previous dental visit
* children suffering from any upper or lower respiratory tract problems
* children with any history of allergy children who currently use any medications

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
anxiety level | salivary cortisol will be assessed by taking saliva samples at baseline, and within 30 minutes of the procedure
  anxiety will be measured by measuring salivary cortisol levels after taking saliva samples

SECONDARY OUTCOMES:
pain perception | immediately after local anesthetic administration
  using Wong-Baker faces pain rating scale Arabic version, the scale has six faces from a happy face for no pain to a crying face for extreme pain, scoring from 0 to 10. Children will be asked to choose the face that expresses their perceived pain intensity
physiological changes(heart rate) | as baseline and 1 minute after local anesthetic administration
  using a finger-type pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Ola Mohamed Abd El-geleel Associate Professor, Study Director — Faculty of Dentistry, Ain Shams University.; Basma Gamal Awad Lecturer, Study Director — Faculty of Dentistry, Ain Shams University.
Locations (1):
- pediatric dentistry and dental public health department, faculty of dentistry, Ain shams university, Cairo, egypt, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Faculty of dentistry Ain Shams University research ethics committee, state that data will not be shared to preserve the confidentiality.